CLINICAL TRIAL: NCT05842109
Title: Clinical Value of ETCOc in the Diagnosis and Treatment of ABO Hemolytic Disease of the Newborn
Brief Title: Clinical Value of ETCOc in the Diagnosis and Treatment of ABO-HDN
Status: Recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: ETCOc in ABO-HDN
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-04

CONDITIONS: ABO Hemolytic Disease of Newborn
Keywords: End tidal carbon monoxide; hyperbilirubinemia; ABO Hemolytic Disease of Newborn
MeSH Terms: conditions — Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ABO HDN: positive in diagnosis of ABO-HDN
- non ABO HDN: negative in diagnosis of ABO-HDN

SUMMARY:
A prospective observational cohort study was designed.

1. Comparing of the clinical indicators between the hemolytic group and the non-hemolytic group,such as End-tidal carbon monoxide corrected for ambient CO(ETCOc),direct antiglobulin test(DAT), the highest total serum bilirubin level and hemoglobin. To explore the role of ETCOc in the diagnosis of neonatal ABO hemolytic disease.
2. Comparing of the clinical indicators between the neonates with IVIG treatment and the neonates without IVIG treatment in ABO hemolytic disease, such as ETCOc,total serum bilirubin level before IVIG treatment and ETCOc,total serum bilirubin level after IVIG treatment.To explore the clinical value of ETCOc in the treatment of ABO hemolytic disease.

DETAILED DESCRIPTION:
A prospective observational cohort study was designed. The participants included in the study are the neonates with hyperbilirubinemia in ABO incompatibility.Because the serological results are not known at the time of enrollment, all the neonates should be suspected hemolysis. According to the serological results,the neonates are divided into two groups, hemolytic group and non-hemolytic group. All the relevant clinical indicators need to be recorded and each neonates needs follow-up.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 35+0 and 41+6 weeks
* birth weight ≥ 2500 grams
* respiratory rate < 60 breaths per minute
* the neonates admitted to the neonatology department for phototherapy because of hyperbilirubinemia that conforms to the guideline of the experts consensus on the management of neonatal hyperbilirubinemia(2014,in China.)
* ABO group incompatibility between the mother and newborn
* the informed consent are obtained.

Exclusion Criteria:

* persistent dyspnea or need for respiratory support
* skin damage or structural deformity around the nasal cavity
* receive intensive care treatment in the neonatal intensive care unit(NICU)
* Severe congenital malformation, chromosomal or genetic abnormality

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: positive in diagnosis of ABO-HDN
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
concentration of ETCOc (end tidal carbon monoxide) | through study completion, planned to be 1.5 year
  ETCOc in ppm

SECONDARY OUTCOMES:
concentration of bilirubin | through study completion, planned to be 1.5 year
  bilirubin in mg/dl
result of DAT | through study completion, planned to be 1.5 year
  DAT result of positive or negtive

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Bao, M.M., Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's hospital School of medicine Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watchko JF. ABO hemolytic disease of the newborn: a need for clarity and consistency in diagnosis. J Perinatol. 2023 Feb;43(2):242-247. doi: 10.1038/s41372-022-01556-6. Epub 2022 Nov 8. PMID 36344813
- [Background] De Winter DP, Hulzebos C, Van 't Oever RM, De Haas M, Verweij EJ, Lopriore E. History and current standard of postnatal management in hemolytic disease of the fetus and newborn. Eur J Pediatr. 2023 Feb;182(2):489-500. doi: 10.1007/s00431-022-04724-0. Epub 2022 Dec 5. PMID 36469119
- [Background] Christensen RD, Bahr TM, Pakdeeto S, Supapannachart S, Zhang H. Perinatal Hemolytic Disorders and Identification Using End Tidal Breath Carbon Monoxide. Curr Pediatr Rev. 2023;19(4):376-387. doi: 10.2174/1573396319666221220095522. PMID 36545740
- [Background] Lozar Krivec J, Lozar Manfreda K, Paro-Panjan D. Clinical Factors Influencing Endogenous Carbon Monoxide Production and Carboxyhemoglobin Levels in Neonates. J Pediatr Hematol Oncol. 2022 Jan 1;44(1):e84-e90. doi: 10.1097/MPH.0000000000002143. PMID 33735151
- [Background] Myle AK, Al-Khattabi GH. Hemolytic Disease of the Newborn: A Review of Current Trends and Prospects. Pediatric Health Med Ther. 2021 Oct 7;12:491-498. doi: 10.2147/PHMT.S327032. eCollection 2021. PMID 34675752
- [Background] Jackson ME, Baker JM. Hemolytic Disease of the Fetus and Newborn: Historical and Current State. Clin Lab Med. 2021 Mar;41(1):133-151. doi: 10.1016/j.cll.2020.10.009. Epub 2020 Dec 24. PMID 33494881
- [Background] Karabulut B, Arcagok BC. A Neglected and Promising Predictor of Severe Hyperbilirubinemia Due to Hemolysis: Carboxyhemoglobin. Fetal Pediatr Pathol. 2020 Apr;39(2):124-131. doi: 10.1080/15513815.2019.1641862. Epub 2019 Jul 19. PMID 31322449
- [Background] Tidmarsh GF, Wong RJ, Stevenson DK. End-tidal carbon monoxide and hemolysis. J Perinatol. 2014 Aug;34(8):577-81. doi: 10.1038/jp.2014.66. Epub 2014 Apr 17. PMID 24743136